CLINICAL TRIAL: NCT04243525
Title: University of Pittsburgh Medical Center (UPMC) Center for Inflammatory Bowel Disease (IBD) Research Registry
Brief Title: Inflammatory Bowel Disease (IBD) Research Registry
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Binion, MD, Professor, University of Pittsburgh
Other Study IDs: STUDY19060285
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Inflamatory Bowel Disease (Crohn's and Ulcerative Colitis)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients seen at the Center for Inflammatory Bowel Disease will be asked to provide their written informed consent (authorization) to allow their identifiable medical record information related to their Inflammatory Bowel Disease to be placed in Center's Research Registry for the purpose of facilitating retrospective research studies directed at Inflammatory Bowel Disease, and the identification and recruitment of potential, eligible subjects for participation in future research studies involving Inflammatory Bowel Disease.

Information obtained from the Inflammatory Bowel Disease Registry will allow a better classification of disease and factors that influence the natural course of disease; which may lead to a better understanding of the pathogenesis of IBD and may permit the development of better therapies and the potential for preventive therapies.

ELIGIBILITY:
Inclusion Criteria:

All patients age 18 and above seeking medical care at the Center for Inflammatory Bowel Diseases Clinic at UPMC

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients-subjects (age 18-100 years old) who are receiving or seeking medical care at the Center for Inflammatory Bowel Diseases Clinic at UPMC
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with IBD | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: David Binion, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States